# **Informed consent form**

**Official Title:** The effect of blood flow restriction training on chronic ankle instability symptoms in sports dance athletes

**Ethical ReviewAcceptance Number: 2023102** 

**Date:** 2023.11.20-2023.12.30

The guarantor: Liu Yang, Wuhan Sports College, Hubei Province, China

**Telephone:** 18935836605

Clinical laboratory; Wuhan Sports Institute Sports Rehabilitation Laboratory and

Wuhan Sports Institute National Fitness Center

### Dear classmates

After passing five tests including Balance Test - Single Leg Stance, Trendelenburg Test, Balance Test - Dynamic Balance Test, Anterior Drawer Test, and Y-Balance Test, two or more tests met the positive test, indicating chronic ankle instability. We have determined that you meet the inclusion criteria for the trial. We invite you to participate in this pilot study, This is an applied study on auxiliary soft tissue release for the treatment of patellofemoral joint pain. This research plan has been approved by the Medical Ethics Committee of Wuhan Sports University. Approval acceptance number: two million twenty-three thousand one hundred and two.

## 1. The purpose of this study

Through experimental observation of exercise intervention (blood flow restriction training combined with low load ankle muscle strength training and balance training) combined with instrument tool therapy (Instrument Soft Tissue Release Technique, IASTM), the intervention effect on ankle function, strength, and joint range of motion of sports dance athletes with ankle instability was observed.

### 2. Inclusion or exclusion criteria for research

Select students majoring in sports dance who have chronic ankle instability and undergo five tests, including balance test, single leg standing, Trendelenburg test, balance test, dynamic balance test, Anterior Drawer test, and Y-Balance test. If two or more tests meet the positive test, it is determined that chronic ankle instability is present, Can be included in the experimental subjects. This experiment has been approved by the Ethics Review Committee of the Medical College of Wuhan Sport University. The specific inclusion and exclusion criteria for subjects are shown in Table 1

**Table 1 Inclusion and Exclusion Criteria** 

| Standard | Inclusion Criteria | Exclusion Criteria |
|---|---|---|
| Age | 118-35 years old | under 18 years old or above 35 years o |
| Course Of | Suffering from chronic ankle instability | Acute ankle injury or no joint injury |
| Disease | symptoms that last for at least 3 months | |

| CAIT score | The CAIT score is 24 points or less. | CAIT score above 24 points |
|---|---|---|
| Functional | Two or more tests tested positive for ankle | Failed ankle function screening |
| screening | joint function screening before the | |
| | experiment | |
| Structural | No structural joint lesions or congenital | Structural lesions or congenital ankle |
| inspection | ankle deformities, | deformities present in the ankle joint |
| Medical | Have not undergone ankle surgery or have | Have undergone ankle surgery or have obvious |
| History | external injuries | injuries or wounds |
| Health | No serious heart, lung, nervous system or | Serious heart, lung, nervous system or other |
| Condition | other systemic diseases | systemic diseases |
| Agree to | Limited athletic ability, unable to complete | Disagree to participate in the study, or inability |
| participate in | research tasks | to understand and comply with the research |
| research | | protocol |

## 3. Research method and process

Methods; 30-45 subjects with ankle instability, restriction or discomfort were selected as observation subjects and randomly divided into blood flow restriction training of the ankle joint combined with IASTM group (n=10-15), blood flow restriction training of the ankle joint alone (n=10-15), and traditional ankle strength training (n=10-15). The intervention was conducted once a week for a total of 4-6 weeks. Cumberland ankle instability assessment, FAAM ankle function assessment score, and ankle range of motion measurements were performed for the three groups at three time points: pre-intervention, post-intervention for the first time, and post-intervention for 4 weeks/6 weeks, respectively. And the ankle strength test was only compared and analyzed at two time points before and after the intervention.

Process: This present study was divided into 3 phases: pre-intervention phase, after the first intervention, and post-intervention phase. In the pre-intervention phase, the researcher will conduct the initial assessment and data statistics of the subjects, including the Cumberland ankle

instability assessment, FAAM ankle function assessment score, and ankle range of motion

measurement. During the intervention phase, subjects in each group will be given a 6-week

exercise intervention with a training frequency of 2 sessions/week of 20-30 minutes each. During

the BFRT exercise, subjects will have a cuff wrapped around the proximal 1/3 of the upper

extremity to achieve the effect of improving muscle strength and endurance by restricting blood

flow, and complete the corresponding ankle training maneuvers (stabilization training,

periarticular ankle muscle group training) in this condition

4. Potential benefits of the study

The experimental exercise intervention may improve the subjects' ankle joint stability and

increase their ankle strength and range of motion.

5. Risks of the study

The BFRT intervention may cause muscle fatigue and thus exacerbate pain, but the intensity

of the exercise is controllable and can be adjusted according to the actual situation

Signature of the subject; Date

Signature of the person in charge of the trial; date